CLINICAL TRIAL: NCT05665348
Title: Randomised, Open-label, Phase II-III Study Evaluating the Benefit of Adding Ipilimumab to the Combination of Atezolizumab and Bevacizumab in Patients With Hepatocellular Carcinoma Receiving First-line Systemic Therapy
Brief Title: Study Evaluating the Benefit of Adding Ipilimumab to the Combination of Atezolizumab and Bevacizumab in Patients With Hepatocellular Carcinoma Receiving First-line Systemic Therapy
Acronym: TRIPLET
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Federation Francophone de Cancerologie Digestive (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FFCD 2101-PRODIGE 81; 2022-501217-31 (EudraCT Number)
Record Dates: First submitted 2022-12-16; First posted 2022-12-27 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: HCC - Hepatocellular Carcinoma; Metastatic Cancer; Metastatic Tumor
Keywords: immunotherapy
MeSH Terms: conditions — Carcinoma, Hepatocellular; Neoplasm Metastasis | interventions — Ipilimumab; atezolizumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DOULET ATEZOLIZUMAB-BEVACIZUMAB (Active Comparator): Standard treatment of HCC by the combination atezolizumab-bevacizumab, 1 cure each 3 weeks during 24 months
  Interventions: Drug: Atezolizumab Injection; Drug: Bevacizumab
- TRIPLET ATEZOLIZUMAB BEVACIZUMAB IPILIMUMAB (Experimental): Standard treatment of HCC by the combination atezolizumab-bevacizumab with addition of ipilimumab for the 4 firsts cures of treatment each 3 weeks, then only treatment by the doublet atezolizumab-bevacizumab each 3 weeks. The total duration of treatment is 24 months.
  Interventions: Drug: Ipilimumab Injection; Drug: Atezolizumab Injection; Drug: Bevacizumab

INTERVENTIONS:
Drug: Ipilimumab Injection — Administration of a combine treatment by atezolizumab and bevacizumab, with addition of ipilimumab for patients enrolled in the experimental arm
  Other Names: Atezolizumab; Bevacizumab
  Arms: TRIPLET ATEZOLIZUMAB BEVACIZUMAB IPILIMUMAB
Drug: Atezolizumab Injection — One of the standard treatment's product for HCC management
Drug: Bevacizumab — One of the standard treatment's product for HCC management

SUMMARY:
TRIPLET HCC is a phase II-III trial that assess the effectivness of addition of ipilimumab to the combination atezolizumab-bevacizumab, on global survival and response to the treatment, for patients with advanced or metastatic hepatocellular carcinoma. The theoretical duration of the study is 5 years. In the scope of this study, each patient will have 2 years of treatment and 2 years of follow-up from their enrollment date.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is one of the most common malignancies and ranks fourth in terms of cancer-related mortality worldwide . Unfortunately, the diagnosis of HCC is often made late in the cure of the disease when the tumour has spread outside the liver parenchyma as portal vein invasion or distant metastases. In the history of HCC patients, a significant proportion will sooner or later face systemic therapies as they are no longer eligible for radical or locoregional therapies. Cytotoxic chemotherapy and hormonal therapies have never shown significant benefit on overall survival (OS) . The first systemic therapy to show a significant beneficial impact on HCC outcome was the tyrosine kinase inhibitor (TKI) sorafenib, an anti-angiogenic agent (AAA) with anti-proliferative properties on HCC . For nearly a decade, all systemic therapies tested in randomised controlled trials as first-line systemic therapy (1L) head-to-head with sorafenib, or as 2L after sorafenib failure have not shown significant benefit. In 2018, Kudo et al. showed that lenvatinib, another TKI with anti-angiogenic properties, was at least equivalent to sorafenib in 1L in the REFLECT non-inferiority trial [5]. Other AAA TKIs with anti-cancer properties on HCC cells have demonstrated efficacy in 2L: regorafenib after progression on sorafenib in 2017 , and cabozantinib after progression on or intolerance to sorafenib in 2018 . In addition, ramucirumab, a monoclonal antibody targeting VEGFR-2, has shown significant benefit in a specific subpopulation of HCC patients with high baseline alpha-fetoprotein levels ≥ 400 ng/ml . However, all these options were strictly palliative with no long-term survivors and lack of potential recovery. Immuno-oncology (IO) approaches have completely revolutionised the paradigm of systemic HCC therapies with nonetheless a significant increase in median OS in IO-based combination strategies, but also the emergence of the possibility of long-term survivors and, for some patients, hope for a complete response and possibly a final cure.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Histologically proven hepatocellular carcinoma (HCC) on biopsy less than two years old. If no histological evidence, a tumour (mandatory) and non-tumour (optional) liver biopsy is required.
* WHO 0 or 1
* HCC not amenable to curative treatment by surgery, thermo-ablation or liver transplantation, or to intra-arterial palliative treatment (IAP) for intermediate BCLC-B HCC.

Advanced (BCLC-C) or intermediate (BCLC-B) HCC after failure or contraindication of the CEL

* Normal Troponin-T
* Patients with controlled cardiovascular disease for at least 6 months
* No clinically evident ascites, no history of clinical ascites, or encephalopathy due to liver failure
* Adequate liver function: AST and ALT ≤ 5 x ULN (upper normal limit), total bilirubin ≤ 35 µM/L, albumin ≥ 28 g/L and Child-Pugh A score (if associated cirrhosis)
* Hematological (hemoglobin > 8.5 g/dL, platelets > 60 G/L, PNN > 1.5 G/L) and renal function (creatinine clearance ≥ 40ml/min according to the appropriate MDRD formula)
* At least one target lesion measurable according to RECIST v1.1 criteria
* Oesophageal endoscopy less than 6 months old. All patients with varicose veins of any grade should be treated with β-blockers prior to initiation of therapy, in the absence of contraindications.
* Women of childbearing potential must agree to use contraception during the trial treatment and for at least 6 months after discontinuation of the experimental treatments. Men who have sex with women of childbearing potential must agree to use contraception during treatment and for at least 6 months after discontinuation of the experimental treatments
* Ability of the patient to understand, sign and date the informed consent form before randomisation
* Patient affiliated to a social security scheme

Exclusion Criteria:

* Patients who have already received systemic therapy for HCC
* Bleeding related to portal hypertension in the last 6 months
* History of abdominal or oesophageal fistula, gastrointestinal perforation or intra-abdominal abscess, diverticulitis or colitis within 6 months prior to randomisation
* Patients on double anti-platelet aggregation therapy
* Patients on chronic non-steroidal anti-inflammatory drugs (except aspirin).
* History of intra-abdominal inflammatory process within 6 months prior to initiation of treatment - including but not limited to - active peptic ulcer, diverticulitis or colitis
* Major surgery or significant traumatic injury within 28 days prior to treatment, abdominal surgery or significant abdominal traumatic injury within 60 days prior to treatment, or the need for major surgery during the therapeutic trial
* Hypersensitivity to any of the study drugs or their excipients
* Allergy to one of the components of Chinese hamster ovary cells.
* Other malignant tumours within the last 2 years, except for carcinoma in situ of the uterus or basal cell or squamous cell skin carcinoma or any other carcinoma in situ, considered curedHistory of severe active life-threatening autoimmune disease
* Interstitial lung disease
* Chronic HBV infection with HBV DNA > 500 IU/ml, infected patients, cirrhotic or not, should be treated with nucleotide/nucleoside analogues.
* Known HIV infection
* Immunosuppression, including subjects with conditions requiring systemic corticosteroid treatment (>10 mg/day prednisone equivalent)
* History of organ transplantation
* Non-healing decaying wound, active ulcer or untreated bone fracture
* Proteinuria ≥ 2+ on urine dipstick if confirmation of 24h proteinuria showing a level ≥ 2 g/24 hours
* Medically uncontrolled hypertension (≥ 150 mm Hg and/or diastolic blood pressure superior to 90 mm Hg)
* History of arterial aneurysm at high risk of bleeding
* Alive attenuated vaccine within 28 days prior to randomisation
* History of pericardial abnormalities possibly immune-related (pericarditis or cardiac tamponade)
* Patient who has received immunotherapy (including anti-CTLA-4, anti-PD-1 or anti-PD-L1 agents) or anti-VEGF antibody therapy
* Patients who has previously received external radiotherapy up to 1 month before the start of the study treatment, or 3 months before the start of the study treatment in case of radio embolization
* Central nervous system metastases
* Active bacterial infection
* Patients with uncontrolled cardiovascular disease
* History of arterial thromboembolic events, including stroke, transient ischemic attack and myocardial infarction, if less than 6 months old and unresolved.
* History of venous thromboembolic disease, if less than 6 months old
* Pregnant or breastfeeding women.
* Person under guardianship, or person deprived of liberty.
* Inability to undergo the medical follow-up of the trial for geographical, social or psychological reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 574 (Estimated)
Dates: Start 2023-03-09 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Objective response of treatment (Phase II) | 24 months after beginning of treatment
  Assess the percentage of patients with an objective response (complete response or partial response) according to the investigator (RECIST v1.1) for both treatments arms,
Overall survival (Phase III) | From randomization until death or last news for alive patients, up to 2 years
  The overall survival is defined as the time to death (whatever the cause) or date of last news

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From randomization until progression, death or last news for alive patients, up to 2 years
  Progression is based on CT-Scan and only radiological progression have to be taking into account. Progression-free survival is defined as the time from randomization to radiological progression or death. Patients alive without progression will be censored at date of last news.
Objective response rate (OR) under treatment (Phase III) | 24 months after beginning of treatment
  Assess the percentage of patients with an objective response (complete response or partial response) according to the investigator (RECIST v1.1) for both treatments

CONTACTS AND LOCATIONS:
Locations (8):
- France (8):
  - Chu Henri Mondor, Créteil
  - Chu Francois Mitterand, Dijon
  - Chu Dupuytren, Limoges
  - Chu La Croix Rousse, Lyon
  - Chu L'Archet, Nice
  - Chu La Pitie Salpetriere, Paris
  - Chu Saint Antoine, Paris
  - Chu Haut Leveque, Pessac